CLINICAL TRIAL: NCT06829524
Title: A Real-World Practical Model of Integrated Management for Chinese Patients with Neuromyelitis Optica Spectrum Disorder (NMOSD) on Satralizumab
Brief Title: HANDLE-a Real World Study on Satralizumab in NMOSD
Status: Not yet recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chao Quan, Professor, Chief Physician, Huashan Hospital
Other Study IDs: KY2024-1393
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Neuromyelitis Optica Spectrum Disorders (NMOSD)
MeSH Terms: conditions — Neuromyelitis Optica | interventions — satralizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Satralizumab treatment group
  Interventions: Drug: Satralizumab

INTERVENTIONS:
Drug: Satralizumab — Satralizumab is the first monoclonal antibody approved for the treatment of NMOSD in China. Currently, there is still a lack of standard patient management pattern for NMOSD. While satralizumab offers the advantage of home administration, there remains a pressing need for optimized patient management.

SUMMARY:
This study is a single-center, retrospective-prospective, non-interventional cohort study to assess the clinical outcomes of Chinese NMOSD patients treated with satralizumab in a real-world patient management model by collecting follow-up data in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have been diagnosed with NMOSD and tested seropositive for AQP4 antibody, ≥ 12 years old;
2. EDSS score ≤ 8.5 at baseline;
3. Patients have experienced ≥ 1 relapse of NMOSD in the last 12 months or ≥ 2 relapses in the last 24 months;
4. Patients should have received or be anticipated to receive satralizumab treatment for at least 12 months;
5. Patients understand the study procedures and sign the informed consent form indicating willingness to participate in the study (for those < 18 years of age, the guardian should sign the informed consent form on behalf of the patient).

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a real-world study and will enroll patients diagnosed with NMOSD who are AQP4-IgG positive and receiving satralizumab in routine clinical practice in China
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients relapse-free at 12 months of treatment with satralizumab | 12 months
Change from baseline in EDSS score at 12 months of treatment with satralizumab | 12 months

SECONDARY OUTCOMES:
Proportion of patients relapse-free at 6 months of treatment with satralizumab | 6 months
Change from baseline in EDSS score at 6 months of treatment with satralizumab | 6 months
Change patterns from baseline in clinical outcome assessments (COAs) at Months 1, 3, 6, and 12 during satralizumab treatment | 1, 3, 6, 12 months
Incidence of AEs and SAEs during satralizumab treatment | 1, 2, 3, 6, 9, 12 months
  Adverse events were coded using MedDRA version 27.1. Adverse events were analyzed in the safety analysis population (all patients who received at least one dose of study treatment) in terms of percentage incidence and as rates by exposure time (number of events per 100 patient-years of exposure and the associated 95% CI) to adjust for any differences in duration of exposure. The severity of adverse events was measured by NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Quan, Doctor, Principal Investigator — Department of Neurology, Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, People's Republic of China; Qiang Dong, Doctor, Study Chair — Department of Neurology, Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, People's Republic of China; Lei Zhou, Study Director — Department of Neurology, Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, People's Republic of China; Wenjuan Huang, Doctor, Study Director — Department of Neurology, Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, People's Republic of China; Jingzi Zhangbao, Doctor, Study Director — Department of Neurology, Huashan Hospital, Shanghai Medical College, Fudan University, Shanghai, People's Republic of China
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No